CLINICAL TRIAL: NCT01405781
Title: Functional and Radiographic Outcomes After Shoulder Surgery
Status: Completed | Type: Observational
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, Robert Tashjian, M.D., University of Utah
Other Study IDs: 46622
Record Dates: First submitted 2011-07-27; First posted 2011-07-29 (Estimated); Last update posted 2025-01-13 (Actual); Status verified 2024-12

CONDITIONS: Shoulder Pain; Osteoarthritis of Glenohumeral Joint; Rotator Cuff Tear Arthropathy
MeSH Terms: conditions — Shoulder Pain; Rotator Cuff Tear Arthropathy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | US Export: No

SUMMARY:
The objective of this study is twofold: First, to determine whether higher levels of pre-operative psychological distress predict worse outcomes after arthroscopic rotator cuff repair; second, to obtain functional outcomes (VAS pain, VAS satisfaction, VAS function, Simple Shoulder Test (SST) and American Shoulder and Elbow Surgeons (ASES) Score), physically examine and perform a radiographic analysis of patients at a minimum of 6 months after reverse total shoulder arthroplasty, total shoulder arthroplasty, arthroscopic scapulothoracic bursectomy, acromioclavicular joint reconstruction and arthroscopic rotator cuff repair.

DETAILED DESCRIPTION:
Clinical outcome studies have been performed in the evaluation of a variety of shoulder pathologies after surgical treatment. Among these disease processes include glenohumeral osteoarthritis, rotator cuff arthropathy, acromioclavicular separations and scapulothoracic bursitis. A variety of outcomes studies have been performed on these pathologies although few have utilized several functional outcome measures. Also with respect to each of these diagnoses, several specific areas of research regarding outcomes assessment have not been investigated.

Glenohumeral osteoarthritis is one of the most common shoulder pathologies treated by orthopedic surgeons. For endstage osteoarthritis, an anatomic total shoulder arthroplasty provides excellent pain relief and functional improvement. In order to perform the replacement, the rotator cuff tendon in the front of the shoulder (subscapularis) needs to be taken down and then repaired at the completion of the case. There are three basic methods of takedown and repair: tenotomy, peel-off and lesser tuberosity osteotomy. The osteotomy has been compared clinically to tenotomy and found to provide a lower rate of subscapularis tears, higher outcome scores and universal healing evaluated using ultrasound and the PENN shoulder score.1 Gerber et al has also evaluated long-term outcomes of total shoulder arthroplasty with lesser osteotomy using the Constant score as a measure of outcomes.2 Unfortunately, many outcome studies evaluating total shoulder arthroplasty utilize the Simple Shoulder Test and the American Shoulder and Elbow Surgeons (ASES) Score which have not been evaluated. Also, osteotomy was performed only utilizing a "fleck" of bone instead of the entire lesser tuberosity. No studies to date have evaluated TSA with an osteotomy of the entire lesser tuberosity.

Reverse total shoulder arthroplasty has shown be a predictable operation for the treatment of rotator cuff arthropathy with clinical improvements in both pain and function at long term. 3,4 Dislocation has been reported between 0% to 9% after reverse total shoulder arthroplasty and has been defined as one of the top three most common complications associated with reverse TSA.3-10 There is considerable debate regarding whether the subscapularis tendon needs repair after reverse TSA. Edwards et al reported a statistically significant reduction in dislocation rates from 9% to 0% with addition of subscapularis repair.10 These results had significant bias with regards to randomization of patients. Similarly, all patients in the non-repair group were at the initial portion of his learning curve. Consequently, the risk for instability is likely lower than reported in his series.

Acromioclavicular joint separations represent one of the most common shoulder injuries accounting for approximately 9% of shoulder girdle injuries.11 Acromioclavicular injuries have been classified with increasing severity from I to VI based upon disruption of the various ligamentous and muscular supports including the acromioclavicular ligaments, coracoclavicular ligaments and deltotrapezial fascia.12 Recommended initial treatment for grade I to III injuries has been nonoperative with reasonable clinical results while initial surgical stabilization has been recommended for higher grade injuries.12-15

A variety of surgical stabilization techniques for acromioclavicular joint separations have been reported including the transfer of the coracoacromial ligament from the acromion to the end of the resected distal clavicle originally described by Weaver and Dunn in 1972.16 A modification of the Weaver-Dunn acromioclavicular reconstruction was subsequently described which included coracoclavicular stabilization with nonabsorbable suture.17 Despite this modification, residual subluxation or dislocation of the acromioclavicular joint has been identified in up to 29% of patients.17 Consequently, alternative constructs have been described including an anatomic reconstruction utilizing a tendon graft which has been shown to have superior biomechanical strength compared to a Weaver-Dunn reconstruction.18

As part of the surgical transition from the modified Weaver-Dunn reconstruction as described by Weinstein et al. to a reconstruction using a tendon graft, augmentation of the coracoclavicular suture fixation with either allograft or autograft tendon as well as performing the coracoacromial ligament transfer has been described.17,19 This differs from the anatomic reconstruction described by Mazzocca et al., as it includes both the transferred coracoacromial ligament and the hamstring graft for stabilization instead of just the graft.11 Coracoclavicular ligament reconstruction with a tendon graft has been reported as a treatment option for failed Weaver-Dunn reconstructions.20,21 Possible benefits of the combined reconstruction include improved construct strength and a vascularized ligament. Drawbacks include increased surgical dissection, increased operating room time and disruption of the coracoacromial arch. With the advances in arthroscopic techniques, acromioclavicular reconstructions utilizing a tendon graft are now being performed arthroscopically which has been described without the addition of coracoacromial ligament transfer.22 Reconstructions without coracoacromial ligament transfers may increase the ease of performing a reconstruction through smaller incisions with arthroscopic assistance. No study has evaluated the clinical effects of adding a coracoacromial ligament transfer to an acromioclavicular joint reconstruction utilizing a coracoclavicular tendon graft.

Scapulothoracic bursitis or "snapping scapula syndrome" is an under-recognized shoulder disorder where the bursal sac between the scapula and chest wall becomes irritated and inflamed. The etiology is overuse causing reactive bursa formation between the scapula and thorax. If conservative measures fail as initial attempts at management, surgical excision of the inflamed bursa with resection of the superior medial angle of the scapula can be performed. The procedure can be performed either arthroscopically or open. A two-portal or three-portal technique can be utilized if performed arthroscopically. Very limited data exists regarding outcomes of two-portal or three-portal techniques with no use of validated patient-based outcome scores.23,24

Rotator cuff tearing is the most common shoulder pathology treated by orthopedic surgeons. Healing rates after rotator cuff repair have varied in the literature from less than 5% to 100% dependent on tear size, age, repair construct and muscle quality.25,26 A variety of methods have been used to repair the tendon. A recent biomechanical study has shown that repair with triple-loaded suture anchors have improved initial biomechanical properties compared to other constructs.27 No clinical data exists on healing after repair with triple loaded anchors or how healing effects function.

ELIGIBILITY:
Inclusion Criteria:

* Patients whose primary presenting complaint of shoulder pain and who then undergo arthroscopic rotator cuff repair performed by the principal investigator for full thickness rotator cuff tear will be eligible for inclusion. All patients who have undergone reverse total shoulder arthroplasty, total shoulder arthroplasty utilizing a lesser tuberosity osteotomy, acromioclavicular joint reconstruction, arthroscopic scapulothoracic bursectomy or arthroscopic rotator cuff repair by the PI (RZT) will also be eligible for inclusion in the study. These will include patients both at the University of Utah as well as the Veteran's Administration Hospital in Salt Lake City. All patients presenting complain of shoulder pain will be given the DRAM survey preoperative and then evaluated a minimum of 6 months postoperative.

Exclusion Criteria:

* All patients who have undergone total shoulder arthroplasty not utilizing a lesser tuberosity osteotomy or who have prior failed rotator cuff repair in the affected shoulder will be excluded.
* All patients who have undergone an open repair of the supraspinatus or infraspinatus rotator cuff tendons will not be eligible.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients whose primary presenting complaint of shoulder pain and who then undergo arthroscopic rotator cuff repair performed by the principal investigator for full thickness rotator cuff tear will be eligible for inclusion. All patients who have undergone reverse total shoulder arthroplasty, total shoulder arthroplasty utilizing a lesser tuberosity osteotomy, acromioclavicular joint reconstruction, arthroscopic scapulothoracic bursectomy or arthroscopic rotator cuff repair by the PI (RZT) will also be eligible for inclusion in the study. These will include patients both at the University of Utah as well as the Veteran's Administration Hospital in Salt Lake City.
Sampling Method: Non-Probability Sample
Enrollment: 1034 (Actual)
Dates: Start 2011-05; Primary Completion 2024-09-13 (Actual); Study Completion 2024-09-13 (Actual)

PRIMARY OUTCOMES:
To determine the outcomes after several different shoulder surgical procedures for varying shoulder problems. | From 6 months

SECONDARY OUTCOMES:
To determine whether higher levels of pre-operative psychological distress predict worse outcomes after arthroscopic rotator cuff repair | from 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Robert z Tashjian, MD, Principal Investigator — University Of Utah Orthopedics Center
Locations (2):
- United States (2):
  - University Of Utah Orthopedics Center, Salt Lake City, Utah
  - Veterans Administration Hospital Salt Lake City, Salt Lake City, Utah